CLINICAL TRIAL: NCT00465699
Title: Evaluation of Topical B12 for the Treatment of Childhood Atopic Dermatitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Spartanburg Regional Healthcare System (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00001369
Record Dates: First submitted 2007-04-23; First posted 2007-04-25 (Estimated); Last update posted 2007-04-25 (Estimated); Status verified 2007-04

CONDITIONS: Eczema
Keywords: Eczema; Pediatric; Vitamin B12
MeSH Terms: conditions — Eczema

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Topical B12 0.07%

SUMMARY:
This study is being done to see in B12 applied to the skin will improve the symptoms of eczema in children compared to a placebo creme

DETAILED DESCRIPTION:
INTRODUCTION: Atopic dermatitis is a prevalent disease process in children, affecting up to 20% of children in the United States. Various treatment options are available to treat atopic dermatitis to include topical emollients, topical steroids, and topical calcineurin inhibitors. Each treatment option has benefits and potential risks. This study was done to determine if topical B12 could be a tolerable and efficacious alternative treatment option in this population.

METHODS: The study was conducted as a placebo-controlled, double-blind, prospective, randomized clinical trial with intraindividual left ⁄ right comparison. Parents were given 2 containers of creams and instructed to apply the Vitamin B12 cream to one side of the body and the placebo cream to the contralateral side according to the randomization scheme.

ELIGIBILITY:
Inclusion Criteria:

* children presenting to the Center for Family Medicine or Regional Pediatrics between the ages of 6 months and 18 years old with atopic dermatitis

Exclusion Criteria:

* unwillingness of parent to consent to study protocol, pregnancy or lactation, eczema with superinfection present, known history of allergy to Vitamin B12 or components of the base cream, topical treatment with corticosteroids in the 4 weeks prior to enrollment

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 50
Dates: Start 2007-04; Study Completion 2007-04 (Estimated)

PRIMARY OUTCOMES:
Reduction in SCORAD at 2 and 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ronald P Januchowski, D.O., Principal Investigator — Spartanburg Regional Healthcare System
Locations (1):
- Center for Family Medicine, Spartanburg, South Carolina, United States

REFERENCES:
- [Background] Stucker M, Pieck C, Stoerb C, Niedner R, Hartung J, Altmeyer P. Topical vitamin B12--a new therapeutic approach in atopic dermatitis-evaluation of efficacy and tolerability in a randomized placebo-controlled multicentre clinical trial. Br J Dermatol. 2004 May;150(5):977-83. doi: 10.1111/j.1365-2133.2004.05866.x. PMID 15149512